CLINICAL TRIAL: NCT04171349
Title: Articaine and Dexmedetomidine - Supplemented Articaine for Arteriovenous Fistula Creation Under Ultrasound- Guided Supraclavicular Block
Brief Title: Articaine vs Dexmedetomidine Supplemented Articaine
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, simon Halim Armanious, Simon Halim, MD S. Armanious, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Articaine
Record Dates: First submitted 2019-11-15; First posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Renal Failure
Keywords: Hemodialysis
MeSH Terms: conditions — Renal Insufficiency | interventions — Carticaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Patients received ultrasound guided supraclavicular block with 40 ml of Articaine hydrochloride 2%
  Interventions: Drug: Articaine
- Group AD (Experimental): Patients received ultrasound guided supraclavicular block with 40 ml articaine 2% mixed with dexmedetomidine (1 µg/kg).
  Interventions: Drug: Articaine; Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Articaine — Vial
Drug: Dexmedetomidine — Vial
  Arms: Group AD

SUMMARY:
The aim of this study to test efficacy of adding dexmedetomidine to articaine on sensory, motor and duration of analgesia during hemodialysis fistula creation under ultrasound guided supraclavicular block

DETAILED DESCRIPTION:
Adult fifty patient with chronic renal failure on hemodialysis, scheduled for arteriovenous fistula creation under ultrasound guided supraclavicular block. Patients were randomly allocated in two group. The articaine group (group A) received 40 ml articaine hydrochloride 2% and articaine-dexmedetomidine group (group AD) received 40 ml. Of articaine 2% mixed with dexmedetomidine (1micogram/kg)

ELIGIBILITY:
Inclusion Criteria:

* adult patient with chronic renal failure on hemodialysis scheduled for radiocephalic fistula creation

Exclusion Criteria:

* Allergy to local anesthetics.
* Infection at the site of needle insertion.
* Those having international normalized ratio more than 1.5.
* Coagulopathy.
* Neuromuscular, or severe hepatic or severe pulmonary disease.
* Those having epilepsy.
* Patients who refused to participate.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Duration of sensory block | 24 hours
  Sensory block time tested by pinprick test measured in minute
Duration of motor block | 24 hours
  Motor block time tested by Bromage scale measured in minutes

SECONDARY OUTCOMES:
Duration of analgesia | 24 hours
  Measured by visual analog scale score 4

OTHER OUTCOMES:
Sedation | 24 hours
  Measured by Ramsay sedation scale score 3

CONTACTS AND LOCATIONS:
Overall Officials: Galal Mo Professor, Doctor, Study Director — Professor
Locations (1):
- Ain Shams University hosptal, Cairo, Abbasya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participants data for all primary and secondary outcome measures will be available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 6 month after study completion
Access Criteria: Data access request will be reviewed by external independent reviewers panal. Request will be required to sign data access

REFERENCES:
- [Derived] Armanious SH, Abdelhameed GA. Articaine and Dexmedetomidine - Supplemented Articaine for Arteriovenous Fistula Creation under Ultrasound-guided Supraclavicular Block. Anesth Essays Res. 2020 Apr-Jun;14(2):248-252. doi: 10.4103/aer.AER_147_19. Epub 2020 Oct 12. PMID 33487824